CLINICAL TRIAL: NCT07039487
Title: EVALUATION OF NEUTROPHIL FLUORESCENCE IN PATIENTS WITH DISSEMINATED INTRAVASCULAR COAGULATION ASSOCIATED WITH SEPTIC SHOCK
Acronym: HEMATOCLOT
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9556; 2024-A02853-44 (Other: ANSM)
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: DISSEMINATED INTRAVASCULAR COAGULATION ASSOCIATED WITH SEPTIC SHOCK

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sampling collection — CBC performed on the background of an EDTA tube, collected routinely allowing neutrophil fluorescence measurements.
  This tube will then be passed over on the automaton for a CBC measurement with leukocyte differentiation.

SUMMARY:
Neutrophil fluorescence could be a reliable and early diagnostic marker of disseminated intravascular coagulation septic DIC, which can be used routinely. The objective of the investigators is to define the optimal threshold of neutrophil fluorescence associated with a sensitivity of at least 90% for the diagnosis of DIC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Patient admitted to intensive care for septic shock
* Patient affiliated to a social security scheme or entitled to it
* Non-opposition by the patient or a relative in the event that the patient is not in a state to express his or her consent or inclusion in an emergency procedure in the event that the patient is not in a state to express his or her opinion and no relative of the patient can be reached.

Exclusion Criteria:

* Dying patient on the day of inclusion
* Cirrhosis Child Pugh C
* Neutropenia (<500 mm3)
* Patient under judicial protection
* Patient under guardianship or curatorship
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to intensive care for septic shock
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Define the optimal threshold for neutrophil fluorescence (measured at admission of the patient to intensive care on a new automaton) associated with a sensitivity of at least 90% for the diagnosis of disseminated intravascular coagulation DIC. | 1 month
  DIC is diagnosed based on the ISTH score (reference diagnosis) on day 2: patients will be considered to have DIC if the score is positive within the first 48 hours after admission to the ICU.
  Neutrophil fluorescence is measured on a new automaton.

SECONDARY OUTCOMES:
To estimate the performance indicators of neutrophil fluorescence measured a new automaton.at admission of the patient to the ICU for all relevant thresholds. | 1 month
  Sensitivity (Se)
To estimate the performance indicators of neutrophil fluorescence measured a new automaton.at admission of the patient to the ICU for all relevant thresholds. | 1 month
  Specificity (Spe)
To estimate the performance indicators of neutrophil fluorescence measured a new automaton.at admission of the patient to the ICU for all relevant thresholds. | 1 month
  Positive Predictive Value (PPV)
To estimate the performance indicators of neutrophil fluorescence measured a new automaton.at admission of the patient to the ICU for all relevant thresholds. | 1 month
  Negative Predictive Value (NPV)
To estimate the performance indicators of neutrophil fluorescence measured a new automaton.at admission of the patient to the ICU for all relevant thresholds. | 1 month
  Positive and Negative Likelihood Ratios of neutrophil fluorescence measured on a new automaton., at dmission to ICU for all relevant thresholds.
To compare the areas under the partial ROC (receiver operating characteristic) curve (for a sensitivity greater than or equal to 90%) illustrating the performance of neutrophil fluorescence measured at the patient's admission to the ICU in the diagnosis | 1 month
  Area under the partial ROC curve (corresponding to a 90% ≥ Se)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Intensive - Réanimation Nouvel Hôpital Civil, Strasbourg, France